CLINICAL TRIAL: NCT05243225
Title: Laparoscopic Versus Open Surgical Management of Post Cholecystectomy Bile Duct Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amir William Samir Fahmy, General Surgery Resident: Amir William Samir Fahmy, Assiut University
Other Study IDs: BDI repair
Record Dates: First submitted 2021-10-26; First posted 2022-02-17 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Bile Duct Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic management of post cholecystectomy bile duct injury.: Under general intubation anaesthesia, trocars are inserted in the abdomen, insufflation by CO2 adhesiolysis is performed to reach the bile duct. Evaluation by intraoperative cholangiogram then according to the site and the size of the injury repair will done. If the injury is small simple repair or repair on T-tube will be done. If the injury is large repair on T-tube or hepaticojejunostomy will be done .If it is a distal injury repair on T-tube or biloenteric shunt will be done .If the injury is proximal biloenteric shunt will be done. Intra-abdominal drains insertion
  Interventions: Procedure: Laparoscopic versus open surgical management of post cholecystectomy bile duct injury
- open surgical management of post cholecystectomy bile duct injury.: Under general intubation anaesthesia, a generous right subcostal incision is performed and could be extended on demand upward to the xiphoid process and/or to the left subcostal area. Thorough dissection and adhesiolysis is performed to reach the bile duct. Evaluation by intraoperative cholangiogram according to the site and the size of the injury repair will be done. If the injury is small simple repair or repair on T-tube will be done . If the injury is large repair on T-tube or hepaticojejunostomy will be done .If it is a distal injury repair on T-tube or biloenteric shunt will be done .If the injury is proximal biloenteric shunt will be done .Intra-abdominal drains insertion.
  Interventions: Procedure: Laparoscopic versus open surgical management of post cholecystectomy bile duct injury

INTERVENTIONS:
Procedure: Laparoscopic versus open surgical management of post cholecystectomy bile duct injury — Comparison between laparoscopic and open surgical management of post cholecystectomy bile duct injury.

SUMMARY:
Comparison between laparoscopic and open surgical management of post cholecystectomy bile duct injury.

DETAILED DESCRIPTION:
Bile duct injury (BDI) post cholecystectomy is an iatrogenic catastrophe associated with significant morbidity , mortality and poor quality of life this is due to the large number of cholecystectomies per year all over the world. Cholecystectomy whether open or laparoscopic is done in large number about 750,000 annually in USA, the incidence of BDI post cholecystectomy is about 0.1-0.2% in open cholecystectomy and 0.4-0.6% in laparoscopic cholecystectomy although the percentage appears small but it still large number about 2100 patients per year. The two most frequent scenarios of BDI may be occurrence of bile leak or bile duct obstruction. Early recognition of iatrogenic bile duct injury is essential to prevent major morbidity by imaging techniques, such as Ultrasound and CT which are extremely valuable during the initial evaluation but MRCP remains the gold standard for diagnosis. ERCP can confirm the presence of biliary injury and provides a means for definitive management. The main aim of surgical treatment is the reconstruction of proper flow of bile to the alimentary tract. Repair of such injuries still remains a challenge due to the variety of size of injury, site of injury if proximal or distal, the severity of injury and the time of presentation after the injury. Repair of such BDI may be done by laparoscopy or by open surgery which still a matter of debate. There are many described techniques should be done by specialized hepatobiliary surgeon from simple repair, repair over T-tube up to hepaticojejunostomy. Despite widespread advances in laparoscopic surgery, laparoscopic repair of post-cholecystectomy bile duct injury (BDI) has rarely been reported related mainly to technical difficulty.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with post cholecystectomy bile duct injuries admitted to surgery department in Asyut University Hospitals and El-Rajhi hospital at the period of the study.
2. Patients fit for surgery.
3. Patients informed consent for study.
4. Patients with signs and symptoms due to Bile duct injury like abdominal pain, jaundice and high liver function parameters

Exclusion Criteria:

1. Unfit cases for laparoscopic surgery.
2. Unfit patients for open surgery.
3. Patients refuse consent to participate in the study.
4. Patients who had previous repair.
5. Patients who present with abdominal sepsis.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with bile duct injury post cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between outcomes of laparoscopic and open surgical management of post cholecystectomy bile duct injury. | Baseline
  Analysis of efficacy of repair in laparoscopic and open surgical management of post cholecystectomy bile duct injury